CLINICAL TRIAL: NCT05593497
Title: Precision Neoadjuvant Therapy for High Risk Localized Prostate Cancer With PTEN Loss
Brief Title: A Single-Arm Phase II Study of Neoadjuvant Intensified Androgen Deprivation (Leuprolide and Abiraterone Acetate) in Combination With AKT Inhibition (Capivasertib) for High-Risk Localized Prostate Cancer With PTEN Loss
Acronym: SNARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-001-21F
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: High-Risk Prostate Cancer
Keywords: veterans; prostate cancer; PTEN protein; prostatectomy; neoadjuvant therapy; abiraterone acetate; capivasertib; leuprolide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — capivasertib; Abiraterone Acetate

STUDY DESIGN:
Intervention Model Description: Eligible patients with high-risk prostate cancer exhibiting <= 10% PTEN staining by IHC will be exposed to a 4-week run-in of iADT, followed by dedicated research biopsy of the tumor to be used for correlative research, then treated with 16 weeks of combined iADT with AKT inhibition (capivasertib). Patients will then undergo radical prostatectomy as standard of care, with assessment of pathological response (pT0 or minimal residual disease) via central pathology review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): neoadjuvant capivasertib combined with androgen receptor pathway therapy (leuprolide + abiraterone) prior to radical prostatectomy
  Interventions: Drug: Capivasertib; Drug: abiraterone acetate

INTERVENTIONS:
Drug: Capivasertib — 400 mg (2 tablets) BID given on an intermittent weekly dosing schedule. Patients will be dosed on Days 1 to 4 in each week (4 days on, 3 days off). Treatment will be given in combination with abiraterone for 16 weeks duration (+/- 1 week for surgery window).
Drug: abiraterone acetate — Administered orally as tablets at a dosage of 1000 mg daily. To be administered with prednisone 5mg po daily.
  Subjects will be on concurrent GNRH agonist therapy (leuprolide, administered as standard of care). Intensified androgen deprivation (iADT) consisting of abiraterone and leuprolide will be administered for a 4 week run-in prior to addition of capivasertib.

SUMMARY:
The purpose of this study is to learn about how an investigational drug intervention completed before doing prostate surgery (specifically, radical prostatectomy with lymph node dissection) may help in treatment of high risk localized prostate cancers that are most resistant to standard treatments. This is a phase II research study. For this study, capivasertib, the study drug, will be taken with intensified androgen deprivation drugs (iADT; abiraterone and leuprolide) prior to radical prostatectomy. This study drug treatment will be evaluated to see if it is effective in shrinking and destroying prostate cancer tumors prior to surgery and to further evaluate its safety prior to prostate cancer surgery.

DETAILED DESCRIPTION:
Prostate cancer is the second leading cause of cancer deaths in men in the United States. Prostate cancer treatment options are historically based on clinical stage, prostate specific antigen (PSA) blood test, and tumor grade. High-risk prostate cancers treated surgically commonly exhibit loss of the phosphatase and tensin homologue (PTEN) tumor suppressor gene, which leads to increased activity of the AKT signaling pathway. PTEN loss is associated with higher rates of prostate cancer recurrence, metastasis, and cancer mortality. Manipulation of androgens and androgen receptor (AR) to reduce mortality has been the focus of prostate cancer systemic therapy for decades; however, PTEN loss is a lead mechanism for prostate cancer resistance to AR directed therapy and development of castrate resistant prostate cancer. Pre-clinical research identified a reciprocal feedback regulation between the PTEN/AKT signaling axis and the Androgen Receptor (AR) signaling axis. Thus, blockade of both pathways may be necessary in tumors with PTEN loss.

This study will change standard localized treatment (radical prostatectomy alone) by conducting a single arm Phase II trial combining intensified androgen deprivation (iADT; abiraterone and leuprolide) with an AKT inhibitor (capivasertib) prior to radical prostatectomy among high-risk localized prostate cancers with PTEN loss. The goal is that early precision treatment of aggressive disease will result minimal residual cancer at the time of prostatectomy, and subsequently improved cancer outcomes.

Eligible patients with high-risk prostate cancer exhibiting 10% PTEN staining by IHC will be exposed to a 4-week run-in of iADT, followed by dedicated research biopsy of the tumor to be used for correlative research, then treated with 16 weeks of combined iADT with AKT inhibition (capivasertib). Patients will then undergo radical prostatectomy as standard of care, with assessment of pathological response (pT0 or minimal residual disease) via central pathology review.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: provision of signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Age greater than or equal to 18 years. Members of all races and ethnic groups will be included.
3. Participants must have histologically confirmed non-metastatic adenocarcinoma of the prostate
4. (a) Any one of the following three high risk features:

   * Gleason sum >7 (ISUP Grade Group >3)
   * Clinical stage T3 (resectable), per AJCC Cancer Staging Manual, 8th ed.
   * PSA > 20 ng/ml oSubjects who meet high risk criteria solely by PSA (i.e., stage <T3 AND Gleason sum less than or equal to 7) must have a progression-free probability after radical prostatectomy that is less than or equal to 50% at 5 years as estimated by the Memorial Sloan Kettering (MSK) pre-radical prostatectomy nomogram: https://www.mskcc.org/nomograms/prostate/pre_op (b) Subjects not meeting high risk criteria that have the following combination may be screened for inclusion:
   * Gleason score 4+3=7 (ISUP Grade Group 3) AND
   * Estimated progression-free probability after radical prostatectomy that is less than or equal to 50% at 5 years by MSK nomogram
5. No definitive evidence of metastasis on nuclear bone scan (required on all subjects)
6. No evidence of lymph nodes > 2 cm in diameter on pelvic CT scan (scan only required in patients with a PSA > 20 ng/ml)
7. Prostatectomy with extended lymph node dissection planned as primary therapy.

   * The subject had a discussion with a clinician about other options, such as radiotherapy, and elected to undergo surgical treatment.
   * The subject has been offered consultation with radiation oncology and declined consultation or radiation treatment, or determined it was not in best medical interest
8. Be willing to provide tissue from a diagnostic biopsy core or excisional biopsy of a tumor lesion obtained up to 6 months/180 days prior to initiation of treatment on Day 1. Subjects for whom samples cannot be provided (e.g., inaccessible or subject safety concern) may submit an older archived specimen only upon agreement from the Sponsor-Investigator.
9. Tumor tissue must be provided for biomarker analysis. PTEN IHC staining must be less than or equal to 10% as determined by the central lab. If insufficient tumor tissue content is provided for analysis, acquisition of additional archived tumor tissue (block and /or slides) for the biomarker analysis is required.
10. Have a performance status of 0 or 1 on the ECOG Performance Scale with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
11. Life expectancy of greater than 10 years per the treating physician.
12. Minimum body weight of 45 kg with minimum Body Mass Index (BMI) of 18.5
13. Non-sterile men who are not totally sexually abstinent (i.e., refraining from heterosexual intercourse during the entire period of risk associated with study interventions) and intend to be sexually active with a women of childbearing potential partner must use a condom upon entering the study and until 16 weeks after the last dose of capivasertib. Contraception should be considered in females' partners of men taking capivasertib who are of childbearing potential
14. Able and willing to swallow and retain oral medication
15. Demonstrate adequate organ function as defined by laboratory parameters including ANC, platelets, hemoglobin, transaminases, albumin, hemoglobin A1C, CrCl or eGFR, PTT and INR (unless anticoagulated, then therapeutic range is acceptable). All screening labs should be performed within 30 days of treatment initiation

Exclusion Criteria:

1. As judged by the investigator, any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant and active bleeding diseases, uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection, cardiac disease) which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
2. Any other disease, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
3. Known to have active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening. Known to have human immunodeficiency virus (HIV) with a CD4+ T-cell count < 350 cells/uL or a history of an acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months. Known to have active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).

   Known history of drug or alcohol abuse within 6 months of screening.
4. Prior prostate cancer treatment including:

   * Anti-androgen therapy including orchiectomy, LHRH therapy, abiraterone, ketoconazole, estrogen therapy (Short-term ADT allowed, less than or equal to 2 months)
   * Radiation (external beam or brachytherapy)
   * Cytotoxic chemotherapy
   * Focal or ablative therapy
   * Any experimental therapy for treatment of prostate cancer.
5. History of another primary malignancy except for malignancy treated with curative intent with no known active disease greater than or equal to 5 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy
6. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive ECGs
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third-degree heart block)
   * Medical history significant for arrhythmia (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted to enter the study
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age, or any concomitant medication known to prolong the QT interval
   * Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or NYHA or Class II to IV heart failure or cardiac ejection fraction measurement of < 50%
   * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade less than or equal to 2
   * Uncontrolled hypotension - systolic blood pressure (SBP) <90 mmHg and/or diastolic blood pressure (DBP) <50 mmHg
   * Uncontrolled hypertension (SBP greater than or equal to 160 mmHg or DBP greater than or equal to 95 mmHg).
   * Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram (or multiple-gated acquisition [MUGA] scan if an echocardiogram cannot be performed or is inconclusive).
7. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   * Patients with diabetes mellitus type 1 or diabetes mellitus type 2 requiring insulin treatment
   * HbA1c greater than or equal to 8.0% (63.9 mmol/mol)
8. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of capivasertib and abiraterone.
9. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
10. Previous allogeneic bone marrow transplant or solid organ transplant
11. Received major surgery within 6 weeks prior to screening, or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study except for prostatectomy; they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
12. Is currently participating and receiving study therapy, or has participated in a study of an investigational agent or study drugs within 30 days or 5 half-lives (whichever is longer) of the first dose of study treatment
13. Has had a prior anti-cancer monoclonal antibody (mAb) within 30 days prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to agents administered more than 30 days earlier.
14. Has had prior chemotherapy, immunotherapy, targeted small molecule therapy, immunosuppressant medication (other than corticosteroids), or radiation therapy within 30 days prior to study Day 1, or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent.

    Note: Subjects with less than or equal to Grade 2 neuropathy are an exception to this criterion and may qualify for the study if ECOG 0-1.

    Note: A longer washout may be required for drugs with a long half-life (e.g., 30 days or 5 half-lives, whichever is longer)
15. Treatment with any of the following:

    * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
    * Potent inhibitors or inducers of CYP3A4 within 2 weeks before the start of study treatment (3 weeks for St John's wort), or sensitive substrates of CYP3A4, CYP2C9 and/or CYP2D6 with a narrow therapeutic window within 1 week before the start of study treatment
    * Drugs known to prolong the QT interval within 5 half-lives of the first dose of study treatment
    * Any concomitant medication that may interfere with abiraterone safety and efficacy based on the prescribing information of abiraterone and local clinical guidelines
16. History of hypersensitivity to active or inactive excipients of capivasertib, abiraterone, or drugs with a similar chemical structure or class.
17. Any restriction or contraindication based on the local prescribing information that would prohibit the use of abiraterone and leuprolide.
18. Is unable to undergo research related biopsy as this is necessary to complete translational study objectives.
19. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response or Minimal Residual Disease (MRD) | 5 months
  No cancer detected on radical prostatectomy specimen, or minimal residual disease 5mm.

SECONDARY OUTCOMES:
Surgical Complications | 5 months + 90 days
  Incidence of Surgical Complications [ Time Frame: 4 months ] Clavien-Dindo Classification of Surgical Complications compared to historical department incidence rates within 90 days after surgery.
ERG Expression and Pathologic Response | 5 months
  No cancer detected on radical prostatectomy specimen, or minimal residual disease 5mm, stratified by normal versus increased ERG expression by immunohistochemistry in prostatectomy specimen

OTHER OUTCOMES:
Treatment related adverse events | 5 months + 90 days
  Grade 3 or higher adverse event (AE) possibly related or related to any of three treatment drugs (capivasertib, abiraterone, leuprolide) per CTCAE v5, evaluated up until 90 days after prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Kopp, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (6):
- United States (6):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No